CLINICAL TRIAL: NCT01667458
Title: F-ACT Trial: Observational Study on Fatigue and Its Evolution During Treatment With Tocilizumab in Patients With Moderate to Severe Rheumatoid Arthritis in Daily Clinical Practice
Brief Title: An Observational Study on Fatigue in Patients With Rheumatoid Arthritis Treated With RoActemra/Actemra (Tocilizumab)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25702
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the presence and evolution of fatigue on treatment with RoActemra/Actemra (tocilizumab) in patients with moderate to severe rheumatoid arthritis who have an inadequate response to at least two DMARDs (one of them methotrexate) or to anti-TNF treatment. Patients initiated on treatment with RoActemra/Actemra (8 mg/kg intravenously every 4 weeks) with or without methotrexate will be followed for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe active rheumatoid arthritis, defined as DAS28 >/= 3.7
* Inadequate clinical response to current treatment with >/= 2 non-biologic DMARDs, 1 of them being methotrexate optimally administered for >/= 3 months, or inadequate clinical response to anti-TNF therapy
* Eligible for RoActemra/Actemra treatment in daily clinical practice
* Absence of evolutive tuberculosis (TB)

Exclusion Criteria:

* Hypersensitivity to tocilizumab or any of the excipients
* Active, severe infections
* Pregnant or lactating women
* Participation in any other interventional study
* Patients with major depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe rheumatoid arthritis with an inadequate response to at least two DMARDs or an inadequate response to anti-TNF treatment, eligible for treatment with RoActemra/Actemra
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Evolution of fatigue: Proportion of patients meeting the Minimally Clinically Important Difference (MCID) for the Visual Analogue Sale VAS Fatigue at Week 16 | 16 months

SECONDARY OUTCOMES:
Fatigue: VAS Fatigue/FACIT Fatigue/Pass Fatigue | 16 months
Disease Activity Score DAS28 | 16 months
Pain: Visual Analogue Scale VAS Pain | 16 months
Functional disability: Health Assessment Questionnaire HAQ | 16 months
Quality of sleep: VAS | 16 months
Anemia: Haemoglobin levels | 16 months
Depression: Beck Depression Inventory (BDI) questionnaire | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Belgium (17):
  - Aalst
  - Assebroek
  - Ath
  - Brussels
  - Dinant
  - Gilly (Charleroi)
  - Kortrijk
  - Lier
  - Mons
  - Namur
  - Roeselare
  - Seraing
  - Sijsele
  - Turnhout
  - Verviers
  - Waremme
  - Westmalle
- Luxembourg, Luxembourg

REFERENCES:
- [Derived] Gossec L, Steinberg G, Rouanet S, Combe B. Fatigue in rheumatoid arthritis: quantitative findings on the efficacy of tocilizumab and on factors associated with fatigue. The French multicentre prospective PEPS Study. Clin Exp Rheumatol. 2015 Sep-Oct;33(5):664-70. Epub 2015 Sep 7. PMID 26344671